CLINICAL TRIAL: NCT00962741
Title: A 2-Part Open-Label Study to Assess the Clinical Benefit and Long-Term Safety of Etanercept in Children and Adolescents With Extended Oligoarticular Juvenile Idiopathic Arthritis, Enthesitis-Related Arthritis, or Psoriatic Arthritis
Brief Title: Study Evaluating Etanercept in 3 Subtypes of Childhood Arthritis
Acronym: CLIPPER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0881A1-3338; B1801014
Record Dates: First submitted 2009-08-13; First posted 2009-08-20 (Estimated); Results first posted 2012-07-19 (Estimated); Last update posted 2014-06-10 (Estimated); Status verified 2014-05

CONDITIONS: Arthritis, Juvenile Idiopathic
MeSH Terms: conditions — Arthritis, Juvenile | interventions — Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Etanercept 0.8 mg/kg QW up to a maximum dose of 50 mg
  Interventions: Drug: Etanercept

INTERVENTIONS:
Drug: Etanercept — Etanercept 0.8 mg/kg QW up to a maximum dose of 50 mg
  Other Names: Enbrel

SUMMARY:
This study will evaluate the effect of etanercept on the clinical benefit, safety, and physical functioning (ability to function in daily life) in children and adolescent subjects with 3 subtypes of childhood arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects with a diagnosis per International League of Associations for Rheumatology (ILAR) criteria of extended oligoarticular juvenile idiopathic arthritis (JIA) between the ages of 2 and 17 years; enthesitis-related arthritis (ERA) between the ages of 12 and 17 years; or psoriatic arthritis (PsA) between the ages of 12 and 17 years.
* >= 2 active joints and the following for the relevant JIA subtype: extended oligoarticular JIA or PsA with a history of intolerance or an unsatisfactory response to a disease modifying antirheumatic drug (DMARD); or ERA with a history of intolerance or an unsatisfactory response to a nonsteroidal anti-inflammatory drug (NSAID) or a DMARD.

Exclusion Criteria:

* Systemic JIA, persistent oligoarticular JIA, polyarticular JIA, or undifferentiated arthritis per ILAR criteria.
* Other rheumatic diseases.
* Active uveitis within 6 months of the baseline visit.
* Any other significant health problem.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 127 (Actual)
Dates: Start 2009-09; Primary Completion 2011-06 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (38):
- Australia (2):
  - Pfizer Investigational Site, Westmead, Sydney, New South Wales
  - Pfizer Investigational Site, Parkville, Melbourne, Victoria
- Belgium (3):
  - Pfizer Investigational Site, Ghent, Belgium
  - Pfizer Investigational Site, Brussels
  - Pfizer Investigational Site, Leuven
- Colombia (3):
  - Pfizer Investigational Site, Barranquilla, Atlántico
  - Pfizer Investigational Site, Bogota, Cundinamarca
  - Pfizer Investigational Site, Bucaramanga, Santander Department
- Czechia (2):
  - Pfizer Investigational Site, Brno
  - Pfizer Investigational Site, Prague
- France (2):
  - Pfizer Investigational Site, Le Kremlin-Bicêtre
  - Pfizer Investigational Site, Paris
- Germany (5):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Bremen
  - Pfizer Investigational Site, Hamburg
  - Pfizer Investigational Site, Hanover
  - Pfizer Investigational Site, Sankt Augustin
- Pfizer Investigational Site, Budapest, Hungary
- Pfizer Investigational Site, Chieti, Italy
- Pfizer Investigational Site, Riga, Latvia
- Pfizer Investigational Site, Vilnius, Lithuania
- Pfizer Investigational Site, Mexico City, Mexico City, Mexico
- Pfizer Investigational Site, Utrecht, Netherlands
- Pfizer Investigational Site, Oslo, Norway
- Poland (4):
  - Pfizer Investigational Site, Krakow, Poland
  - Pfizer Investigational Site, Wroclaw, Poland
  - Pfizer Investigational Site, Bydgoszcz
  - Pfizer Investigational Site, Warsaw
- Russia (2):
  - Pfizer Investigational Site, Moscow
  - Pfizer Investigational Site, Saint Petersburg
- Serbia (2):
  - Pfizer Investigational Site, Belgrade, Serbia
  - Pfizer Investigational Site, Niš
- Slovakia (2):
  - Pfizer Investigational Site, Košice
  - Pfizer Investigational Site, Piešťany
- Pfizer Investigational Site, Ljubljana, Slovenia
- Spain (3):
  - Pfizer Investigational Site, Esplugues de Llobregat, Barcelona
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Valencia, Valencia

REFERENCES:
- [Derived] Vojinovic J, Foeldvari I, Dehoorne J, Panaviene V, Susic G, Horneff G, Stanevicha V, Kobusinska K, Zuber Z, Dobrzyniecka B, Akikusa J, Avcin T, Borlenghi C, Arthur E, Tatulych SY, Zang C, Tsekouras V, Vlahos B, Martini A, Ruperto N. Ten-year safety and clinical benefit from open-label etanercept treatment in children and young adults with juvenile idiopathic arthritis. Rheumatology (Oxford). 2024 Jan 4;63(1):140-148. doi: 10.1093/rheumatology/kead183. PMID 37140539
- [Derived] Foeldvari I, Constantin T, Vojinovic J, Horneff G, Chasnyk V, Dehoorne J, Panaviene V, Susic G, Stanevicha V, Kobusinska K, Zuber Z, Dobrzyniecka B, Nikishina I, Bader-Meunier B, Breda L, Dolezalova P, Job-Deslandre C, Rumba-Rozenfelde I, Wulffraat N, Pedersen RD, Bukowski JF, Vlahos B, Martini A, Ruperto N; Paediatric Rheumatology International Trials Organisation (PRINTO). Etanercept treatment for extended oligoarticular juvenile idiopathic arthritis, enthesitis-related arthritis, or psoriatic arthritis: 6-year efficacy and safety data from an open-label trial. Arthritis Res Ther. 2019 May 23;21(1):125. doi: 10.1186/s13075-019-1916-9. PMID 31122296
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=0881A1-3338&StudyName=Study%20Evaluating%20Etanercept%20in%203%20Subtypes%20of%20Childhood%20Arthritis

RESULTS

PARTICIPANT FLOW:
Groups:
- Etanercept: Etanercept was administered 0.8 milligram/kilogram (mg/kg) up to a maximum dose of 50 mg once weekly subcutaneously for 96 weeks.
Period: Overall Study
Arm/Group | Etanercept
Started | 127
Completed | 119
Not Completed | 8
Not completed — Failed to return | 3
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 1
Not completed — Lack of Efficacy | 1
Not completed — drug ineffective+prohibited drug taken | 1

BASELINE CHARACTERISTICS:
Groups:
- Etanercept: Etanercept was administered 0.8 mg/kg up to a maximum dose of 50 mg once weekly subcutaneously for 96 weeks.
Arm/Group | Etanercept
Number analyzed (Participants) | 127
Age, Continuous [Mean (Standard Deviation); unit: Years] | 11.70 (4.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72
  Male | 55

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an American College of Rheumatology Pediatric 30 (ACR Pedi 30) Response at Week 12
Description: ACR Pedi 30 response: greater than or equal to (>=) 30% improvement from baseline in 3 of 6 criteria with worsening > 30% in no more than 1 of 6 criteria: 1) physician's global assessment of disease activity, 2) parent/patient global assessment of arthritis pain, 3) childhood health assessment questionnaire (CHAQ) 4) number of active joints 5) number of joints with limited range of motion and 6) C-reactive protein.
Time Frame: Week 12
Population: Modified Intent-to-Treat (mITT) population included all participants who received at least 1 dose of the study medication. Here 'N' (Number of participants analyzed) signified those participants who were evaluable for this measure at week 12.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 123
Percentage of participants | 88.6 [81.6 to 93.6]

2. Secondary Outcome: Percentage of Participants With an ACR Pedi 30 Response
Description: ACR Pedi 30 response: >= 30% improvement from baseline in 3 of 6 criteria with worsening > 30% in no more than 1 of 6 criteria: 1) physician's global assessment of disease activity, 2) parent/patient global assessment of arthritis pain, 3) CHAQ 4) number of active joints 5) number of joints with limited range of motion and 6) C-reactive protein.
Time Frame: Week 4, Week 8, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: mITT population included all participants who received at least 1 dose of the study medication. Data are presented for Part 1 (up to 12 weeks) and Part 2 (up to 96 weeks).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 127
Percentage of participants
  Week 4 (N = 126) | 71.4 [62.7 to 79.1]
  Week 8 (N = 121) | 88.4 [81.3 to 93.5]
  Week 12 (N = 123) | 88.6 [81.6 to 93.6]
  Week 24 (N = 122) | 94.3 [88.5 to 97.7]
  Week 36 (N = 120) | 95.8 [90.5 to 98.6]
  Week 48 (N = 119) | 94.1 [88.3 to 97.6]
  Week 60 (N = 116) | 95.7 [90.2 to 98.6]
  Week 72 (N = 114) | 96.5 [91.3 to 99.0]
  Week 84 (N = 113) | 93.8 [87.7 to 97.5]
  Week 96 (N = 108) | 99.1 [94.9 to 100]

3. Secondary Outcome: Percentage of Participants With an ACR Pedi 30 Response: Extended Oligoarticular Juvenile Idiopathic Arthritis (eoJIA) Sub-population
Description: as for outcome 2
Time Frame: Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: eoJIA: participants with arthritis affecting 1 to 4 joints during the first 6 months of the disease and had progressed to affect more than 4 joints after the first 6 months of disease. Data are presented for Part 1 (up to 12 weeks) and Part 2 (up to 96 weeks).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 60
Percentage of participants
  Week 4 (N = 59) | 67.8 [54.4 to 79.4]
  Week 8 (N = 56) | 87.5 [75.9 to 94.8]
  Week 12 (N = 58) | 89.7 [78.8 to 96.1]
  Week 24 (N = 58) | 94.8 [85.6 to 98.9]
  Week 36 (N = 57) | 94.7 [85.4 to 98.9]
  Week 48 (N = 57) | 96.5 [87.9 to 99.6]
  Week 60 (N = 56) | 98.2 [90.4 to 100]
  Week 72 (N = 55) | 98.2 [90.3 to 100]
  Week 84 (N = 55) | 98.2 [90.3 to 100]
  Week 96 (N = 53) | 100 [93.3 to 100]

4. Secondary Outcome: Percentage of Participants With an ACR Pedi 30 Response: Enthesitis-Related Arthritis (ERA) Sub-population
Description: ACR Pedi 30 response: >= 30% improvement from baseline in 3 of 6 criteria with worsening > 30% in no more than 1 of 6 criteria: 1) physician's global assessment of disease activity, 2) parent/patient global assessment of arthritis pain, 3) CHAQ 4) number of active joints 5) number of joints with limited range of motion and 6) C-reactive protein. Data are presented for Part 1 (up to 12 weeks) and Part 2 (up to 96 weeks).
Time Frame: Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: ERA:participants with arthritis(Ar) or(/)enthesitis,any 2:sacroiliac joint tenderness/inflammatory(Ifm)lumbosacral pain history;ankylosing spondylitis,ERA,sacroiliitis with Ifm bowel disease,Reiter's syndrome history;human leukocyte antigen;Ar in male>6years;acute anterior uveitis(AAU)/AAU first-degree relative.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 38
Percentage of participants
  Week 4 (N = 38) | 84.2 [68.7 to 94.0]
  Week 8 (N = 36) | 91.7 [77.5 to 98.2]
  Week 12 (N = 36) | 83.3 [67.2 to 93.6]
  Week 24 (N = 36) | 91.7 [77.5 to 98.2]
  Week 36 (N = 35) | 97.1 [85.1 to 99.9]
  Week 48 (N = 34) | 91.2 [76.3 to 98.1]
  Week 60 (N = 33) | 90.9 [75.7 to 98.1]
  Week 72 (N = 32) | 93.8 [79.2 to 99.2]
  Week 84 (N = 31) | 90.3 [74.2 to 98.0]
  Week 96 (N = 30) | 100 [88.4 to 100]

5. Secondary Outcome: Percentage of Participants With an ACR Pedi 30 Response: Psoriatic Arthritis (PsA) Sub-population
Description: as for outcome 2
Time Frame: Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: PsA: participants with arthritis and psoriasis, or arthritis plus at least 2 of the following: 1) dactylitis; 2) nail pitting or onycholysis; 3) psoriasis in a first-degree relative. Data are presented for Part 1 (up to 12 weeks) and Part 2 (up to 96 weeks).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 29
Percentage of participants
  Week 4 (N = 29) | 62.1 [42.3 to 79.3]
  Week 8 (N = 29) | 86.2 [68.3 to 96.1]
  Week 12 (N = 29) | 93.1 [77.2 to 99.2]
  Week 24 (N = 28) | 96.4 [81.7 to 99.9]
  Week 36 (N = 28) | 96.4 [81.7 to 99.9]
  Week 48 (N = 28) | 92.9 [76.5 to 99.1]
  Week 60 (N = 27) | 96.3 [81.0 to 99.9]
  Week 72 (N = 27) | 96.3 [81.0 to 99.9]
  Week 84 (N = 27) | 88.9 [70.8 to 97.6]
  Week 96 (N = 25) | 96.0 [79.6 to 99.9]

6. Secondary Outcome: Percentage of Participants With an ACR Pedi 50 Response
Description: ACR Pedi 50 response: >= 50% improvement from baseline in 3 of 6 criteria with worsening > 30% in no more than 1 of 6 criteria: 1) physician's global assessment of disease activity, 2) parent/patient global assessment of disease activity, 3) CHAQ 4) number of active joints 5) number of joints with limited range of motion and 6) C-reactive protein at each visit.
Time Frame: Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 127
Percentage of participants
  Week 4 (N = 125) | 51.2 [42.1 to 60.2]
  Week 8 (N = 121) | 76.9 [68.3 to 84.0]
  Week 12 (N = 122) | 81.1 [73.1 to 87.7]
  Week 24 (N = 122) | 88.5 [81.5 to 93.6]
  Week 36 (N = 120) | 88.3 [81.2 to 93.5]
  Week 48 (N = 119) | 93.3 [87.2 to 97.1]
  Week 60 (N = 116) | 92.2 [85.8 to 96.4]
  Week 72 (N = 114) | 93.9 [87.8 to 97.5]
  Week 84 (N = 113) | 91.2 [84.3 to 95.7]
  Week 96 (N = 108) | 98.1 [93.5 to 99.8]

7. Secondary Outcome: Percentage of Participants With an ACR Pedi 50 Response: eoJIA Sub-population
Description: as for outcome 6
Time Frame: Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 60
Percentage of participants
  Week 4 (N = 58) | 51.7 [38.2 to 65.0]
  Week 8 (N = 56) | 75.0 [61.6 to 85.6]
  Week 12 (N = 58) | 79.3 [66.6 to 88.8]
  Week 24 (N = 58) | 86.2 [74.6 to 93.9]
  Week 36 (N = 57) | 91.2 [80.7 to 97.1]
  Week 48 (N = 57) | 94.7 [85.4 to 98.9]
  Week 60 (N = 56) | 92.9 [82.7 to 98.0]
  Week 72 (N = 55) | 96.4 [87.5 to 99.6]
  Week 84 (N = 55) | 96.4 [87.5 to 99.6]
  Week 96 (N = 53) | 100 [93.3 to 100]

8. Secondary Outcome: Percentage of Participants With an ACR Pedi 50 Response: ERA Sub-population
Description: as for outcome 6
Time Frame: Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: ERA: participants with Ar/enthesitis,any 2:sacroiliac joint tenderness/Ifm lumbosacral pain history; ankylosing spondylitis,ERA,sacroiliitis with Ifm bowel disease,Reiter's syndrome history;human leukocyte antigen;Ar in male>6years;AAU/AAU in first-degree relative. Data are presented for Part 1 (up to 12 weeks) and Part 2 (up to 96 weeks).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 38
Percentage of participants
  Week 4 (N = 38) | 63.2 [46.0 to 78.2]
  Week 8 (N = 36) | 86.1 [70.5 to 95.3]
  Week 12 (N = 35) | 80.0 [63.1 to 91.6]
  Week 24 (N = 36) | 86.1 [70.5 to 95.3]
  Week 36 (N = 35) | 82.9 [66.4 to 93.4]
  Week 48 (N = 34) | 91.2 [76.3 to 98.1]
  Week 60 (N = 33) | 87.9 [71.8 to 96.6]
  Week 72 (N = 32) | 90.6 [75.0 to 98.0]
  Week 84 (N = 31) | 83.9 [66.3 to 94.5]
  Week 96 (N = 30) | 96.7 [82.8 to 99.9]

9. Secondary Outcome: Percentage of Participants With an ACR Pedi 50 Response: PsA Sub-population
Description: as for outcome 6
Time Frame: Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 29
Percentage of participants
  Week 4 (N = 29) | 34.5 [17.9 to 54.3]
  Week 8 (N = 29) | 69.0 [49.2 to 84.7]
  Week 12 (N = 29) | 86.2 [68.3 to 96.1]
  Week 24 (N = 28) | 96.4 [81.7 to 99.9]
  Week 36 (N = 28) | 89.3 [71.8 to 97.7]
  Week 48 (N = 28) | 92.9 [76.5 to 99.1]
  Week 60 (N = 27) | 96.3 [81.0 to 99.9]
  Week 72 (N = 27) | 92.6 [75.7 to 99.1]
  Week 84 (N = 27) | 88.9 [70.8 to 97.6]
  Week 96 (N = 25) | 96.0 [79.6 to 99.9]

10. Secondary Outcome: Percentage of Participants With an ACR Pedi 70 Response
Description: ACR Pedi 70 response: >= 70% improvement from baseline in 3 of 6 criteria with worsening > 30% in no more than 1 of 6 criteria: 1) physician's global assessment of disease activity, 2) parent/patient global assessment of disease activity, 3) CHAQ 4) number of active joints 5) number of joints with limited range of motion and 6) C-reactive protein at each visit.
Time Frame: Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 127
Percentage of participants
  Week 4 (N = 126) | 26.2 [18.8 to 34.8]
  Week 8 (N = 121) | 47.1 [38.0 to 56.4]
  Week 12 (N = 122) | 61.5 [52.2 to 70.1]
  Week 24 (N = 122) | 71.3 [62.4 to 79.1]
  Week 36 (N = 120) | 73.3 [64.5 to 81.0]
  Week 48 (N = 119) | 79.8 [71.5 to 86.6]
  Week 60 (N = 115) | 81.7 [73.5 to 88.3]
  Week 72 (N = 114) | 84.2 [76.2 to 90.4]
  Week 84 (N = 113) | 87.6 [80.1 to 93.1]
  Week 96 (N = 108) | 92.6 [85.9 to 96.7]

11. Secondary Outcome: Percentage of Participants With an ACR Pedi 70 Response: eoJIA Sub-population
Description: as for outcome 10
Time Frame: Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 60
Percentage of participants
  Week 4 (N = 59) | 28.8 [17.8 to 42.1]
  Week 8 (N = 56) | 51.8 [38.0 to 65.3]
  Week 12 (N = 58) | 63.8 [50.1 to 76.0]
  Week 24 (N = 58) | 70.7 [57.3 to 81.9]
  Week 36 (N = 57) | 75.4 [62.2 to 85.9]
  Week 48 (N = 57) | 77.2 [64.2 to 87.3]
  Week 60 (N = 55) | 80.0 [67.0 to 89.6]
  Week 72 (N = 55) | 85.5 [73.3 to 93.5]
  Week 84 (N = 55) | 90.9 [80.0 to 97.0]
  Week 96 (N = 53) | 94.3 [84.3 to 98.8]

12. Secondary Outcome: Percentage of Participants With an ACR Pedi 70 Response: ERA Sub-population
Description: as for outcome 10
Time Frame: Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 38
Percentage of participants
  Week 4 (N = 38) | 28.9 [15.4 to 45.9]
  Week 8 (N = 36) | 52.8 [35.5 to 69.6]
  Week 12 (N = 35) | 71.4 [53.7 to 85.4]
  Week 24 (N = 36) | 80.6 [64.0 to 91.8]
  Week 36 (N = 35) | 77.1 [59.9 to 89.6]
  Week 48 (N = 34) | 85.3 [68.9 to 95.0]
  Week 60 (N = 33) | 81.8 [64.5 to 93.0]
  Week 72 (N = 32) | 81.3 [63.6 to 92.8]
  Week 84 (N = 31) | 80.6 [62.5 to 92.5]
  Week 96 (N = 30) | 86.7 [69.3 to 96.2]

13. Secondary Outcome: Percentage of Participants With an ACR Pedi 70 Response: PsA Sub-population
Description: as for outcome 10
Time Frame: Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 29
Percentage of participants
  Week 4 (N = 29) | 17.2 [5.8 to 35.8]
  Week 8 (N = 29) | 31.0 [15.3 to 50.8]
  Week 12 (N = 29) | 44.8 [26.4 to 64.3]
  Week 24 (N = 28) | 60.7 [40.6 to 78.5]
  Week 36 (N = 28) | 64.3 [44.1 to 81.4]
  Week 48 (N = 28) | 78.6 [59.0 to 91.7]
  Week 60 (N = 27) | 85.2 [66.3 to 95.8]
  Week 72 (N = 27) | 85.2 [66.3 to 95.8]
  Week 84 (N = 27) | 88.9 [70.8 to 97.6]
  Week 96 (N = 25) | 96.0 [79.6 to 99.9]

14. Secondary Outcome: Percentage of Participants With an ACR Pedi 90 Response
Description: ACR Pedi 90 response: >= 90% improvement from baseline in 3 of 6 criteria with worsening > 30% in no more than 1 of 6 criteria: 1) physician's global assessment of disease activity, 2) parent/patient global assessment of disease activity, 3) CHAQ 4) number of active joints 5) number of joints with limited range of motion and 6) C-reactive protein at each visit.
Time Frame: Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 127
Percentage of participants
  Week 4 (N = 126) | 6.3 [2.8 to 12.1]
  Week 8 (N = 121) | 14.9 [9.1 to 22.5]
  Week 12 (N = 121) | 29.8 [21.8 to 38.7]
  Week 24 (N = 122) | 43.4 [34.5 to 52.7]
  Week 36 (N = 120) | 47.5 [38.3 to 56.8]
  Week 48 (N = 119) | 50.4 [41.1 to 59.7]
  Week 60 (N = 115) | 53.0 [43.5 to 62.4]
  Week 72 (N = 113) | 60.2 [50.5 to 69.3]
  Week 84 (N = 113) | 64.6 [55.0 to 73.4]
  Week 96 (N = 107) | 65.4 [55.6 to 74.4]

15. Secondary Outcome: Percentage of Participants With an ACR Pedi 90 Response:eoJIA Sub-population
Description: as for outcome 14
Time Frame: Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 60
Percentage of participants
  Week 4 (N = 59) | 6.8 [1.9 to 16.5]
  Week 8 (N = 56) | 16.1 [7.6 to 28.3]
  Week 12 (N = 58) | 27.6 [16.7 to 40.9]
  Week 24 (N = 58) | 53.4 [39.9 to 66.7]
  Week 36 (N = 57) | 49.1 [35.6 to 62.7]
  Week 48 (N = 57) | 52.6 [39.0 to 66.0]
  Week 60 (N = 55) | 52.7 [38.8 to 66.3]
  Week 72 (N = 54) | 61.1 [46.9 to 74.1]
  Week 84 (N = 55) | 67.3 [53.3 to 79.3]
  Week 96 (N = 53) | 62.3 [47.9 to 75.2]

16. Secondary Outcome: Percentage of Participants With an ACR Pedi 90 Response: ERA Sub-population
Description: as for outcome 14
Time Frame: Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 38
Percentage of participants
  Week 4 (N = 38) | 10.5 [2.9 to 24.8]
  Week 8 (N = 36) | 22.2 [10.1 to 39.2]
  Week 12 (N = 35) | 45.7 [28.8 to 63.4]
  Week 24 (N = 36) | 41.7 [25.5 to 59.2]
  Week 36 (N = 35) | 48.6 [31.4 to 66.0]
  Week 48 (N = 34) | 50.0 [32.4 to 67.6]
  Week 60 (N = 33) | 57.6 [39.2 to 74.5]
  Week 72 (N = 32) | 71.9 [53.3 to 86.3]
  Week 84 (N = 31) | 64.5 [45.4 to 80.8]
  Week 96 (N = 30) | 66.7 [47.2 to 82.7]

17. Secondary Outcome: Percentage of Participants With an ACR Pedi 90 Response: PsA Sub-population
Description: as for outcome 14
Time Frame: Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 29
Percentage of participants
  Week 4 (N = 29) | 0.0 [0.0 to 11.9]
  Week 8 (N = 29) | 3.4 [0.1 to 17.8]
  Week 12 (N = 28) | 14.3 [4.0 to 32.7]
  Week 24 (N = 28) | 25.0 [10.7 to 44.9]
  Week 36 (N = 28) | 42.9 [24.5 to 62.8]
  Week 48 (N = 28) | 46.4 [27.5 to 66.1]
  Week 60 (N = 27) | 48.1 [28.7 to 68.1]
  Week 72 (N = 27) | 44.4 [25.5 to 64.7]
  Week 84 (N = 27) | 59.3 [38.8 to 77.6]
  Week 96 (N = 24) | 70.8 [48.3 to 87.4]

18. Secondary Outcome: Percentage of Participants With an ACR Pedi 100 Response
Description: ACR Pedi 100 response: 100% improvement from baseline in 3 of 6 criteria with worsening > 30% in no more than 1 of 6 criteria: 1) physician's global assessment of disease activity, 2) parent/patient global assessment of disease activity, 3) CHAQ 4) number of active joints 5) number of joints with limited range of motion and 6) C-reactive protein at each visit.
Time Frame: Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 127
Percentage of participants
  Week 4 (N = 126) | 3.2 [0.9 to 7.9]
  Week 8 (N = 121) | 6.6 [2.9 to 12.6]
  Week 12 (N = 122) | 23.0 [15.8 to 31.4]
  Week 24 (N = 122) | 33.6 [25.3 to 42.7]
  Week 36 (N = 120) | 36.7 [28.1 to 45.9]
  Week 48 (N = 119) | 40.3 [31.4 to 49.7]
  Week 60 (N = 114) | 42.1 [32.9 to 51.7]
  Week 72 (N = 113) | 49.6 [40.0 to 59.1]
  Week 84 (N = 112) | 55.4 [45.7 to 64.8]
  Week 96 (N = 107) | 54.2 [44.3 to 63.9]

19. Secondary Outcome: Percentage of Participants With an ACR Pedi 100 Response: eoJIA Sub-population
Description: as for outcome 18
Time Frame: Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 60
Percentage of participants
  Week 4 (N = 59) | 6.8 [1.9 to 16.5]
  Week 8 (N = 56) | 8.9 [3.0 to 19.6]
  Week 12 (N = 58) | 20.7 [11.2 to 33.4]
  Week 24 (N = 58) | 39.7 [27.0 to 53.4]
  Week 36 (N = 57) | 42.1 [29.1 to 55.9]
  Week 48 (N = 57) | 47.4 [34.0 to 61.0]
  Week 60 (N = 55) | 47.3 [33.7 to 61.2]
  Week 72 (N = 54) | 51.9 [37.8 to 65.7]
  Week 84 (N = 55) | 60.0 [45.9 to 73.0]
  Week 96 (N = 53) | 54.7 [40.4 to 68.4]

20. Secondary Outcome: Percentage of Participants With an ACR Pedi 100 Response: ERA Sub-population
Description: as for outcome 18
Time Frame: Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 38
Percentage of participants
  Week 4 (N = 38) | 0.0 [0.0 to 9.3]
  Week 8 (N = 36) | 5.6 [0.7 to 18.7]
  Week 12 (N = 35) | 34.3 [19.1 to 52.2]
  Week 24 (N = 36) | 36.1 [20.8 to 53.8]
  Week 36 (N = 35) | 34.3 [19.1 to 52.2]
  Week 48 (N = 34) | 32.4 [17.4 to 50.5]
  Week 60 (N = 33) | 42.4 [25.5 to 60.8]
  Week 72 (N = 32) | 59.4 [40.6 to 76.3]
  Week 84 (N = 31) | 54.8 [36.0 to 72.7]
  Week 96 (N = 30) | 50.0 [31.3 to 68.7]

21. Secondary Outcome: Percentage of Participants With an ACR Pedi 100 Response: PsA Sub-population
Description: as for outcome 18
Time Frame: Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 29
Percentage of participants
  Week 4 (N = 29) | 0.0 [0.0 to 11.9]
  Week 8 (N = 29) | 3.4 [0.1 to 17.8]
  Week 12 (N = 29) | 13.8 [3.9 to 31.7]
  Week 24 (N = 28) | 17.9 [6.1 to 36.9]
  Week 36 (N = 28) | 28.6 [13.2 to 48.7]
  Week 48 (N = 28) | 35.7 [18.6 to 55.9]
  Week 60 (N = 26) | 30.8 [14.3 to 51.8]
  Week 72 (N = 27) | 33.3 [16.5 to 54.0]
  Week 84 (N = 26) | 46.2 [36.6 to 66.6]
  Week 96 (N = 24) | 58.3 [36.6 to 77.9]

22. Secondary Outcome: Physician's Global Assessment (PGA) of Disease Activity
Description: PGA of Disease Activity was measured on a 21-circle Visual Analog Scale (VAS) ranging from 0 to 10, with 0 = no disease activity and 10= Maximum disease activity.
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 127
Units on a scale
  Baseline (N = 127) | 5.02 (1.75)
  Week 4 (N = 126) | 2.78 (1.78)
  Week 8 (N = 121) | 2.00 (1.55)
  Week 12 (N = 123) | 1.50 (1.30)
  Week 24 (N = 122) | 1.15 (1.22)
  Week 36 (N = 120) | 1.05 (1.17)
  Week 48 (N = 119) | 1.03 (1.19)
  Week 60 (N = 116) | 0.88 (0.99)
  Week 72 (N = 113) | 0.78 (0.97)
  Week 84 (N = 113) | 0.78 (1.04)
  Week 96 (N = 108) | 0.62 (0.79)

23. Secondary Outcome: Physician's Global Assessment (PGA) of Disease Activity: eoJIA Sub-population
Description: as for outcome 22
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: eoJIA: participants with arthritis affecting 1 to 4 joints during the first 6 months of the disease that progressed to affect more than 4 joints after the first 6 months of disease. Data are presented for Part 1 (up to 12 weeks) and Part 2 (up to 96 weeks).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 60
Units on a scale
  Baseline (N = 60) | 4.96 (1.76)
  Week 4 (N = 59) | 2.73 (1.80)
  Week 8 (N = 56) | 1.80 (1.62)
  Week 12 (N = 58) | 1.40 (1.30)
  Week 24 (N = 58) | 1.03 (1.34)
  Week 36 (N = 57) | 0.89 (1.25)
  Week 48 (N = 57) | 0.88 (1.20)
  Week 60 (N = 56) | 0.83 (1.06)
  Week 72 (N = 54) | 0.72 (0.99)
  Week 84 (N = 55) | 0.60 (0.86)
  Week 96 (N = 53) | 0.59 (0.81)

24. Secondary Outcome: Physician's Global Assessment (PGA) of Disease Activity: ERA Sub-population
Description: as for outcome 22
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 38
Units on a scale
  Baseline (N = 38) | 5.39 (1.94)
  Week 4 (N = 38) | 2.71 (1.94)
  Week 8 (N = 36) | 2.19 (1.50)
  Week 12 (N = 36) | 1.53 (1.34)
  Week 24 (N = 36) | 1.32 (1.12)
  Week 36 (N = 35) | 1.21 (1.10)
  Week 48 (N = 34) | 1.16 (1.14)
  Week 60 (N = 33) | 0.80 (0.87)
  Week 72 (N = 32) | 0.78 (0.98)
  Week 84 (N = 31) | 0.84 (1.09)
  Week 96 (N = 30) | 0.62 (0.67)

25. Secondary Outcome: Physician's Global Assessment (PGA) of Disease Activity: PsA Sub-population
Description: as for outcome 22
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 29
Units on a scale
  Baseline (N = 29) | 4.66 (1.42)
  Week 4 (N = 29) | 2.98 (1.56)
  Week 8 (N = 29) | 2.14 (1.49)
  Week 12 (N = 29) | 1.69 (1.28)
  Week 24 (N = 28) | 1.18 (1.06)
  Week 36 (N = 28) | 1.20 (1.09)
  Week 48 (N = 28) | 1.18 (1.22)
  Week 60 (N = 27) | 1.06 (0.99)
  Week 72 (N = 27) | 0.89 (0.93)
  Week 84 (N = 27) | 1.07 (1.25)
  Week 96 (N = 25) | 0.66 (0.90)

26. Secondary Outcome: Patient/Parent Global Assessment
Description: Patient/Parent Global Assessment was assessed by the participant's parent using a 21-circle VAS ranging from 0 to 10, with 0 = very well and 10 = very poor.
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 127
Units on a scale
  Baseline (N = 127) | 4.96 (2.33)
  Week 4 (N = 126) | 3.22 (2.23)
  Week 8 (N = 121) | 2.79 (2.10)
  Week 12 (N = 123) | 2.21 (1.84)
  Week 24 (N = 122) | 1.79 (1.75)
  Week 36 (N = 120) | 1.74 (1.97)
  Week 48 (N = 119) | 1.65 (1.88)
  Week 60 (N = 116) | 1.33 (1.56)
  Week 72 (N = 114) | 1.29 (1.63)
  Week 84 (N = 113) | 1.17 (1.56)
  Week 96 (N = 109) | 0.97 (1.31)

27. Secondary Outcome: Patient/Parent Global Assessment: eoJIA Sub-population
Description: as for outcome 26
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 60
Units on a scale
  Baseline (N = 60) | 4.82 (2.44)
  Week 4 (N = 59) | 2.82 (2.11)
  Week 8 (N = 56) | 2.38 (2.02)
  Week 12 (N = 58) | 1.97 (1.81)
  Week 24 (N = 58) | 1.51 (1.69)
  Week 36 (N = 57) | 1.56 (2.07)
  Week 48 (N = 57) | 1.32 (1.82)
  Week 60 (N = 56) | 1.29 (1.54)
  Week 72 (N = 55) | 1.17 (1.55)
  Week 84 (N = 55) | 0.90 (1.21)
  Week 96 (N = 54) | 1.00 (1.43)

28. Secondary Outcome: Patient/Parent Global Assessment: ERA Sub-population
Description: as for outcome 26
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 38
Units on a scale
  Baseline (N = 38) | 5.43 (2.26)
  Week 4 (N = 38) | 3.62 (2.43)
  Week 8 (N = 36) | 3.19 (2.26)
  Week 12 (N = 36) | 2.56 (2.13)
  Week 24 (N = 36) | 2.26 (2.03)
  Week 36 (N = 35) | 2.04 (2.05)
  Week 48 (N = 34) | 2.07 (2.14)
  Week 60 (N = 33) | 1.39 (1.74)
  Week 72 (N = 32) | 1.39 (1.80)
  Week 84 (N = 31) | 1.29 (1.60)
  Week 96 (N = 30) | 0.93 (1.19)

29. Secondary Outcome: Patient/Parent Global Assessment: PsA Sub-population
Description: as for outcome 26
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 29
Units on a scale
  Baseline (N = 29) | 4.62 (2.17)
  Week 4 (N = 29) | 3.50 (2.14)
  Week 8 (N = 29) | 3.10 (1.97)
  Week 12 (N = 29) | 2.26 (1.46)
  Week 24 (N = 28) | 1.75 (1.38)
  Week 36 (N = 28) | 1.73 (1.64)
  Week 48 (N = 28) | 1.82 (1.61)
  Week 60 (N = 27) | 1.33 (1.42)
  Week 72 (N = 27) | 1.39 (1.64)
  Week 84 (N = 27) | 1.59 (2.05)
  Week 96 (N = 25) | 0.96 (1.22)

30. Secondary Outcome: Number of Active Joints
Description: Active joints: Joints that were swollen or, in absence of swelling, joints with limited motion with pain and/or tenderness. Joints were coded as: 0= no swelling, limitation of motion, or pain and/or tenderness on motion; 1= any swelling, limitation of motion, or pain and/or tenderness on motion; JR= joint replacement; NE= not evaluable. Total number of active joints= 73*(total number of active joints with counts > 0)/number of non-missing active joints. JR and NE were treated as missing. If > 36 active joint counts were missing, total number of active joints was defined as missing.
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Joints
Arm/Group | Etanercept
Number analyzed (Participants) | 127
Joints
  Baseline (N = 127) | 6.74 (4.59)
  Week 4 (N = 126) | 3.17 (3.32)
  Week 8 (N = 121) | 2.07 (2.67)
  Week 12 (N = 123) | 1.72 (2.52)
  Week 24 (N = 122) | 1.16 (2.06)
  Week 36 (N = 120) | 0.99 (1.86)
  Week 48 (N = 119) | 0.88 (1.92)
  Week 60 (N = 116) | 0.87 (1.94)
  Week 72 (N = 114) | 0.77 (1.97)
  Week 84 (N = 113) | 0.81 (2.20)
  Week 96 (N = 109) | 0.61 (2.06)

31. Secondary Outcome: Number of Active Joints: eoJIA Sub-population
Description: as for outcome 30
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: Joints
Arm/Group | Etanercept
Number analyzed (Participants) | 60
Joints
  Baseline (N = 60) | 7.58 (5.09)
  Week 4 (N = 59) | 3.95 (3.75)
  Week 8 (N = 56) | 2.46 (2.70)
  Week 12 (N = 58) | 2.07 (2.77)
  Week 24 (N = 58) | 1.34 (2.29)
  Week 36 (N = 57) | 1.14 (1.97)
  Week 48 (N = 57) | 1.00 (1.60)
  Week 60 (N = 56) | 0.98 (1.63)
  Week 72 (N = 55) | 0.73 (1.21)
  Week 84 (N = 55) | 0.65 (1.16)
  Week 96 (N = 54) | 0.50 (0.89)

32. Secondary Outcome: Number of Active Joints: ERA Sub-population
Description: as for outcome 30
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Joints
Arm/Group | Etanercept
Number analyzed (Participants) | 38
Joints
  Baseline (N = 38) | 5.21 (3.57)
  Week 4 (N = 38) | 2.40 (2.62)
  Week 8 (N = 36) | 1.47 (2.25)
  Week 12 (N = 36) | 1.08 (1.57)
  Week 24 (N = 36) | 0.78 (1.07)
  Week 36 (N = 35) | 0.74 (1.29)
  Week 48 (N = 34) | 0.68 (1.09)
  Week 60 (N = 33) | 0.48 (0.94)
  Week 72 (N = 32) | 0.59 (1.21)
  Week 84 (N = 31) | 0.68 (1.19)
  Week 96 (N = 30) | 0.50 (0.94)

33. Secondary Outcome: Number of Active Joints: PsA Sub-population
Description: as for outcome 30
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Joints
Arm/Group | Etanercept
Number analyzed (Participants) | 29
Joints
  Baseline (N = 29) | 7.00 (4.33)
  Week 4 (N = 29) | 2.59 (2.92)
  Week 8 (N = 29) | 2.07 (3.05)
  Week 12 (N = 29) | 1.79 (2.86)
  Week 24 (N = 28) | 1.25 (2.47)
  Week 36 (N = 28) | 1.00 (2.21)
  Week 48 (N = 28) | 0.89 (3.03)
  Week 60 (N = 27) | 1.11 (3.11)
  Week 72 (N = 27) | 1.08 (3.45)
  Week 84 (N = 27) | 1.30 (4.02)
  Week 96 (N = 25) | 0.96 (4.00)

34. Secondary Outcome: Number of Joints With Limitation of Motion
Description: The joints were assessed and coded as: 0= no limitation of motion; 1= any limitation of motion; JR= joint replacement; NE= not evaluable. Total number of joints with limitation of motion: 69*(total number of joints with counts of limitation of motion > 0)/number of non-missing limitation of motions. JR and NE were treated as missing. If > 34 counts of limitation of motion were missing, total number of joints with limitation of motion was defined as missing.
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Joints
Arm/Group | Etanercept
Number analyzed (Participants) | 127
Joints
  Baseline (N = 127) | 5.72 (4.22)
  Week 4 (N = 126) | 3.20 (3.27)
  Week 8 (N = 121) | 2.26 (3.41)
  Week 12 (N = 123) | 1.62 (2.31)
  Week 24 (N = 122) | 1.43 (2.03)
  Week 36 (N = 120) | 1.39 (2.13)
  Week 48 (N = 119) | 1.26 (2.51)
  Week 60 (N = 116) | 1.41 (2.98)
  Week 72 (N = 114) | 1.13 (2.36)
  Week 84 (N = 113) | 1.41 (3.05)
  Week 96 (N = 109) | 1.06 (2.71)

35. Secondary Outcome: Number of Joints With Limitation of Motion: eoJIA Sub-population
Description: as for outcome 34
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: Joints
Arm/Group | Etanercept
Number analyzed (Participants) | 60
Joints
  Baseline (N = 60) | 6.33 (4.37)
  Week 4 (N = 59) | 3.12 (2.74)
  Week 8 (N = 56) | 2.23 (3.47)
  Week 12 (N = 58) | 1.78 (2.25)
  Week 24 (N = 58) | 1.40 (1.77)
  Week 36 (N = 57) | 1.16 (1.54)
  Week 48 (N = 57) | 1.05 (1.63)
  Week 60 (N = 56) | 1.36 (2.56)
  Week 72 (N = 55) | 0.89 (1.58)
  Week 84 (N = 55) | 0.98 (2.08)
  Week 96 (N = 54) | 0.74 (1.22)

36. Secondary Outcome: Number of Joints With Limitation of Motion: ERA Sub-population
Description: as for outcome 34
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Joints
Arm/Group | Etanercept
Number analyzed (Participants) | 38
Joints
  Baseline (N = 38) | 4.84 (4.00)
  Week 4 (N = 38) | 2.98 (3.73)
  Week 8 (N = 36) | 2.28 (3.59)
  Week 12 (N = 36) | 1.58 (2.94)
  Week 24 (N = 36) | 1.53 (2.80)
  Week 36 (N = 35) | 1.55 (2.69)
  Week 48 (N = 34) | 1.53 (2.88)
  Week 60 (N = 33) | 1.36 (3.26)
  Week 72 (N = 32) | 1.19 (2.09)
  Week 84 (N = 31) | 1.68 (3.17)
  Week 96 (N = 30) | 1.33 (2.89)

37. Secondary Outcome: Number of Joints With Limitation of Motion: PsA Sub-population
Description: as for outcome 34
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Joints
Arm/Group | Etanercept
Number analyzed (Participants) | 29
Joints
  Baseline (N = 29) | 5.62 (4.10)
  Week 4 (N = 29) | 3.66 (3.66)
  Week 8 (N = 29) | 2.28 (3.15)
  Week 12 (N = 29) | 1.34 (1.40)
  Week 24 (N = 28) | 1.36 (1.31)
  Week 36 (N = 28) | 1.64 (2.39)
  Week 48 (N = 28) | 1.36 (3.42)
  Week 60 (N = 27) | 1.56 (3.51)
  Week 72 (N = 27) | 1.56 (3.68)
  Week 84 (N = 27) | 1.96 (4.34)
  Week 96 (N = 25) | 1.40 (4.39)

38. Secondary Outcome: C-reactive Protein (CRP)
Description: The test for CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation. A decrease in the level of CRP indicates reduction in inflammation and therefore improvement.
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/Liter (mg/L)
Arm/Group | Etanercept
Number analyzed (Participants) | 127
mg/Liter (mg/L)
  Baseline (N = 127) | 8.26 (14.70)
  Week 4 (N = 125) | 3.29 (7.85)
  Week 8 (N = 121) | 2.32 (3.92)
  Week 12 (N = 120) | 2.47 (7.19)
  Week 24 (N = 120) | 3.54 (10.72)
  Week 36 (N = 119) | 2.81 (5.75)
  Week 48 (N = 117) | 2.04 (3.94)
  Week 60 (N = 110) | 2.16 (4.87)
  Week 72 (N = 111) | 2.26 (4.01)
  Week 84 (N = 109) | 3.98 (12.51)
  Week 96 (N = 103) | 2.76 (5.27)

39. Secondary Outcome: C-reactive Protein (CRP): eoJIA Sub-population
Description: as for outcome 38
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Etanercept
Number analyzed (Participants) | 60
mg/L
  Baseline (N = 60) | 6.27 (10.59)
  Week 4 (N = 58) | 3.45 (7.79)
  Week 8 (N = 56) | 2.66 (5.05)
  Week 12 (N = 58) | 3.36 (10.07)
  Week 24 (N = 56) | 5.26 (15.34)
  Week 36 (N = 57) | 3.25 (6.56)
  Week 48 (N = 55) | 1.93 (4.20)
  Week 60 (N = 55) | 2.76 (6.52)
  Week 72 (N = 55) | 2.42 (4.28)
  Week 84 (N = 54) | 3.94 (9.13)
  Week 96 (N = 52) | 3.34 (6.62)

40. Secondary Outcome: C-reactive Protein (CRP): ERA Sub-population
Description: as for outcome 38
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Etanercept
Number analyzed (Participants) | 38
mg/L
  Baseline (N = 38) | 15.27 (21.52)
  Week 4 (N = 38) | 4.37 (10.36)
  Week 8 (N = 36) | 2.53 (3.30)
  Week 12 (N = 34) | 1.87 (2.84)
  Week 24 (N = 36) | 1.96 (2.04)
  Week 36 (N = 35) | 3.24 (6.41)
  Week 48 (N = 34) | 2.79 (4.89)
  Week 60 (N = 30) | 1.99 (2.84)
  Week 72 (N = 30) | 2.12 (4.03)
  Week 84 (N = 29) | 6.36 (20.81)
  Week 96 (N = 27) | 2.68 (4.10)

41. Secondary Outcome: C-reactive Protein (CRP): PsA Sub-population
Description: as for outcome 38
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Etanercept
Number analyzed (Participants) | 29
mg/L
  Baseline (N = 29) | 3.19 (4.71)
  Week 4 (N = 29) | 1.58 (1.73)
  Week 8 (N = 29) | 1.41 (0.98)
  Week 12 (N = 28) | 1.36 (0.75)
  Week 24 (N = 28) | 2.11 (3.16)
  Week 36 (N = 27) | 1.31 (0.81)
  Week 48 (N = 28) | 1.35 (0.97)
  Week 60 (N = 25) | 1.04 (0.12)
  Week 72 (N = 26) | 2.08 (3.51)
  Week 84 (N = 26) | 1.44 (0.97)
  Week 96 (N = 24) | 1.58 (2.18)

42. Secondary Outcome: Pain Assessment
Description: Pain Assessment was assessed by the participant's parent using a 21-circle VAS ranging from 0 to 10, with 0 = no pain and 10 = very severe pain.
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 127
Units on a scale
  Baseline (N = 127) | 5.06 (2.52)
  Week 4 (N = 126) | 3.12 (2.25)
  Week 8 (N = 121) | 2.58 (2.10)
  Week 12 (N = 123) | 2.02 (1.89)
  Week 24 (N = 122) | 1.64 (1.74)
  Week 36 (N = 120) | 1.63 (1.94)
  Week 48 (N = 119) | 1.51 (1.81)
  Week 60 (N = 116) | 1.18 (1.46)
  Week 72 (N = 114) | 1.14 (1.62)
  Week 84 (N = 112) | 1.13 (1.67)
  Week 96 (N = 108) | 0.91 (1.42)

43. Secondary Outcome: Pain Assessment: eoJIA Sub-population
Description: as for outcome 42
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 60
Units on a scale
  Baseline (N = 60) | 4.81 (2.56)
  Week 4 (N = 59) | 2.64 (2.09)
  Week 8 (N = 56) | 2.12 (1.97)
  Week 12 (N = 58) | 1.69 (1.77)
  Week 24 (N = 58) | 1.27 (1.66)
  Week 36 (N = 57) | 1.43 (1.98)
  Week 48 (N = 57) | 1.19 (1.77)
  Week 60 (N = 56) | 1.19 (1.38)
  Week 72 (N = 55) | 1.01 (1.52)
  Week 84 (N = 54) | 0.91 (1.50)
  Week 96 (N = 53) | 0.97 (1.52)

44. Secondary Outcome: Pain Assessment: ERA Sub-population
Description: as for outcome 42
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 38
Units on a scale
  Baseline (N = 38) | 5.76 (2.51)
  Week 4 (N = 38) | 3.82 (2.59)
  Week 8 (N = 36) | 3.13 (2.42)
  Week 12 (N = 36) | 2.54 (2.18)
  Week 24 (N = 36) | 2.28 (1.89)
  Week 36 (N = 35) | 1.87 (2.07)
  Week 48 (N = 34) | 1.78 (1.72)
  Week 60 (N = 33) | 1.17 (1.69)
  Week 72 (N = 32) | 1.17 (1.69)
  Week 84 (N = 31) | 1.08 (1.34)
  Week 96 (N = 30) | 0.87 (1.21)

45. Secondary Outcome: Pain Assessment: PsA Sub-population
Description: as for outcome 42
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 29
Units on a scale
  Baseline (N = 29) | 4.64 (2.31)
  Week 4 (N = 29) | 3.19 (1.91)
  Week 8 (N = 29) | 2.81 (1.74)
  Week 12 (N = 29) | 2.03 (1.65)
  Week 24 (N = 28) | 1.61 (1.51)
  Week 36 (N = 28) | 1.71 (1.67)
  Week 48 (N = 28) | 1.82 (1.95)
  Week 60 (N = 27) | 1.19 (1.35)
  Week 72 (N = 27) | 1.37 (1.74)
  Week 84 (N = 27) | 1.61 (2.20)
  Week 96 (N = 25) | 0.84 (1.48)

46. Secondary Outcome: Duration of Morning Stiffness
Description: Duration of morning stiffness was defined as the time elapsed when participant woke up in the morning and was able to resume normal activities without stiffness in minutes (If none was present = 0; If morning stiffness was continuing at the time of assessment or was unusual compared to the recent past, average of duration of stiffness over the past 3 days was reported; If stiffness persisted the entire day, 1440 minutes was recorded).
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Etanercept
Number analyzed (Participants) | 127
Minutes
  Baseline (N = 127) | 73.50 (100.61)
  Week 4 (N = 126) | 29.86 (60.00)
  Week 8 (N = 121) | 25.02 (75.32)
  Week 12 (N = 123) | 13.29 (41.20)
  Week 24 (N = 122) | 8.83 (23.41)
  Week 36 (N = 120) | 6.76 (24.41)
  Week 48 (N = 119) | 6.01 (23.94)
  Week 60 (N = 116) | 7.28 (30.28)
  Week 72 (N = 113) | 8.98 (30.67)
  Week 84 (N = 112) | 8.40 (32.38)
  Week 96 (N = 109) | 5.76 (21.70)

47. Secondary Outcome: Duration of Morning Stiffness: eoJIA Sub-population
Description: as for outcome 46
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Etanercept
Number analyzed (Participants) | 60
Minutes
  Baseline (N = 60) | 72.78 (97.24)
  Week 4 (N = 59) | 20.46 (47.37)
  Week 8 (N = 56) | 20.18 (70.70)
  Week 12 (N = 58) | 9.05 (24.52)
  Week 24 (N = 58) | 5.72 (18.85)
  Week 36 (N = 57) | 2.49 (9.35)
  Week 48 (N = 57) | 2.19 (6.61)
  Week 60 (N = 56) | 2.41 (7.32)
  Week 72 (N = 54) | 3.89 (15.16)
  Week 84 (N = 55) | 2.64 (8.97)
  Week 96 (N = 54) | 2.37 (12.42)

48. Secondary Outcome: Duration of Morning Stiffness: ERA Sub-population
Description: as for outcome 46
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Etanercept
Number analyzed (Participants) | 38
Minutes
  Baseline (N = 38) | 89.29 (128.94)
  Week 4 (N = 38) | 49.34 (78.73)
  Week 8 (N = 36) | 44.03 (102.65)
  Week 12 (N = 36) | 25.69 (67.57)
  Week 24 (N = 36) | 15.69 (28.87)
  Week 36 (N = 35) | 17.17 (41.01)
  Week 48 (N = 34) | 13.38 (36.88)
  Week 60 (N = 33) | 14.09 (42.21)
  Week 72 (N = 32) | 16.25 (42.12)
  Week 84 (N = 30) | 12.70 (36.16)
  Week 96 (N = 30) | 10.67 (28.31)

49. Secondary Outcome: Duration of Morning Stiffness: PsA Sub-population
Description: as for outcome 46
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Etanercept
Number analyzed (Participants) | 29
Minutes
  Baseline (N = 29) | 54.31 (54.16)
  Week 4 (N = 29) | 23.45 (49.86)
  Week 8 (N = 29) | 10.79 (24.55)
  Week 12 (N = 29) | 6.38 (13.42)
  Week 24 (N = 28) | 6.43 (23.17)
  Week 36 (N = 28) | 2.43 (11.33)
  Week 48 (N = 28) | 4.82 (25.51)
  Week 60 (N = 27) | 9.07 (40.43)
  Week 72 (N = 27) | 10.56 (36.70)
  Week 84 (N = 27) | 15.37 (52.05)
  Week 96 (N = 25) | 7.20 (27.43)

50. Secondary Outcome: Percentage of Participants With Inactive Disease Per Wallace 2004 Definition
Description: Inactive disease was defined as no joints with active arthritis, a normal CRP, and a PGA of Disease Activity of 0 on a 21-circle VAS.
Time Frame: Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 127
Percentage of participants
  Week 4 (N = 126) | 2.4
  Week 8 (N = 121) | 2.5
  Week 12 (N = 123) | 12.2
  Week 24 (N = 121) | 24.8
  Week 36 (N = 120) | 25.0
  Week 48 (N = 118) | 29.7
  Week 60 (N = 113) | 33.6
  Week 72 (N = 111) | 36.0
  Week 84 (N = 110) | 34.5
  Week 96 (N = 106) | 34.0

51. Secondary Outcome: Percentage of Participants With Inactive Disease Per Wallace 2004 Definition: eoJIA Sub-population
Description: as for outcome 50
Time Frame: Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 60
Percentage of participants
  Week 4 (N = 59) | 5.1
  Week 8 (N = 56) | 3.6
  Week 12 (N = 58) | 12.1
  Week 24 (N = 57) | 29.8
  Week 36 (N = 57) | 35.1
  Week 48 (N = 56) | 37.5
  Week 60 (N = 56) | 48.2
  Week 72 (N = 54) | 46.3
  Week 84 (N = 54) | 44.4
  Week 96 (N = 53) | 37.7

52. Secondary Outcome: Percentage of Participants With Inactive Disease Per Wallace 2004 Definition: ERA Sub-population
Description: as for outcome 50
Time Frame: Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: ERA:participants with Ar/enthesitis,any 2:sacroiliac joint tenderness/Ifm lumbosacral pain history;ankylosing spondylitis,ERA,sacroiliitis with Ifm bowel disease,Reiter's syndrome history;humanleukocyte antigen;Ar in male>6years;AAU/AAU in first-degree relative. Data are presented for Part 1 (up to 12 weeks) and Part 2 (up to 96 weeks).
Measure: Number; unit: Percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 38
Percentage of participants
  Week 4 (N = 38) | 0.0
  Week 8 (N = 36) | 2.8
  Week 12 (N = 36) | 16.7
  Week 24 (N = 36) | 25.0
  Week 36 (N = 35) | 14.3
  Week 48 (N = 34) | 23.5
  Week 60 (N = 30) | 23.3
  Week 72 (N = 30) | 33.3
  Week 84 (N = 29) | 27.6
  Week 96 (N = 28) | 28.6

53. Secondary Outcome: Percentage of Participants With Inactive Disease Per Wallace 2004 Definition: PsA Sub-population
Description: as for outcome 50
Time Frame: Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 29
Percentage of participants
  Week 4 (N = 29) | 0.0
  Week 8 (N = 29) | 0.0
  Week 12 (N = 29) | 6.9
  Week 24 (N = 28) | 14.3
  Week 36 (N = 28) | 17.9
  Week 48 (N = 28) | 21.4
  Week 60 (N = 27) | 14.8
  Week 72 (N=27) | 18.5
  Week 84 (N = 27) | 22.2
  Week 96 (N = 25) | 32.0

54. Secondary Outcome: Childhood Health Assessment Questionnaire (CHAQ) Score
Description: CHAQ: parent-administered, valid assessment of functional disability, discomfort in pediatrics with rheumatic diseases. Parents report participants's ability to perform activities in 8 domains: dressing, arising, eating, walking,hygiene, each,grip,common activities distributed in total of 30 items.Each item is scored on 4-point Likert scale: 0=no difficulty;1=some difficulty;2=much difficulty;3=unable to do. Highest score reported for domain is score for that domain.Overall score = sum of domain scores divided by number of domains answered. Total score: 0=no difficulty to 3=extreme difficulty.
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 127
Units on a scale
  Baseline (N = 127) | 0.80 (0.63)
  Week 4 (N = 126) | 0.54 (0.55)
  Week 8 (N = 121) | 0.42 (0.45)
  Week 12 (N = 123) | 0.32 (0.40)
  Week 24 (N = 122) | 0.28 (0.39)
  Week 36 (N = 120) | 0.23 (0.39)
  Week 48 (N = 119) | 0.24 (0.41)
  Week 60 (N = 116) | 0.20 (0.37)
  Week 72 (N = 114) | 0.17 (0.32)
  Week 84 (N = 113) | 0.17 (0.35)
  Week 96 (N = 109) | 0.16 (0.35)

55. Secondary Outcome: Childhood Health Assessment Questionnaire (CHAQ) Score: eoJIA Sub-population
Description: as for outcome 54
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 60
Units on a scale
  Baseline (N = 60) | 0.90 (0.68)
  Week 4 (N = 59) | 0.64 (0.60)
  Week 8 (N = 56) | 0.50 (0.54)
  Week 12 (N = 58) | 0.40 (0.48)
  Week 24 (N = 58) | 0.31 (0.43)
  Week 36 (N = 57) | 0.26 (0.46)
  Week 48 (N = 57) | 0.27 (0.48)
  Week 60 (N = 56) | 0.25 (0.45)
  Week 72 (N = 55) | 0.21 (0.37)
  Week 84 (N = 55) | 0.21 (0.41)
  Week 96 (N = 54) | 0.20 (0.40)

56. Secondary Outcome: Childhood Health Assessment Questionnaire (CHAQ) Score: ERA Sub-population
Description: as for outcome 54
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: ERA: participants with Ar /enthesitis,any 2:sacroiliac joint tenderness/Ifm lumbosacral pain history; ankylosing spondylitis,ERA,sacroiliitis with Ifm bowel disease,Reiter's syndrome history;human leukocyte antigen;Ar in male>6years;AAU/AAU in first-degree relative. Data are presented for Part 1 (up to 12 weeks) and Part 2 (up to 96 weeks).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 38
Units on a scale
  Baseline (N = 38) | 0.72 (0.51)
  Week 4 (N = 38) | 0.48 (0.56)
  Week 8 (N = 36) | 0.40 (0.34)
  Week 12 (N = 36) | 0.23 (0.27)
  Week 24 (N = 36) | 0.27 (0.38)
  Week 36 (N = 35) | 0.20 (0.32)
  Week 48 (N = 34) | 0.18 (0.28)
  Week 60 (N = 33) | 0.17 (0.29)
  Week 72 (N = 32) | 0.13 (0.27)
  Week 84 (N = 31) | 0.10 (0.22)
  Week 96 (N = 30) | 0.08 (0.21)

57. Secondary Outcome: Childhood Health Assessment Questionnaire (CHAQ) Score: PsA Sub-population
Description: as for outcome 54
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 29
Units on a scale
  Baseline (N = 29) | 0.68 (0.63)
  Week 4 (N = 29) | 0.42 (0.41)
  Week 8 (N = 29) | 0.30 (0.34)
  Week 12 (N = 29) | 0.29 (0.35)
  Week 24 (N = 28) | 0.26 (0.32)
  Week 36 (N = 28) | 0.21 (0.32)
  Week 48 (N = 28) | 0.24 (0.38)
  Week 60 (N = 27) | 0.13 (0.25)
  Week 72 (N = 27) | 0.15 (0.29)
  Week 84 (N = 27) | 0.18 (0.35)
  Week 96 (N = 25) | 0.18 (0.36)

58. Other Pre Specified Outcome: Tender Entheseal Assessment for ERA Sub-population
Description: Tender entheseal assessment: Entheses were assessed and coded as: 1= any tenderness, 0= no tenderness, NE= not evaluable. Total number of tender entheses: 66*(total number of tender entheses with counts > 0)/number of non-missing tender entheses. If > 33 tender entheseal counts were missing, total number of tender entheses was defined as missing.
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Tender entheses
Arm/Group | Etanercept
Number analyzed (Participants) | 38
Tender entheses
  Baseline (N = 38) | 5.87 (9.42)
  Week 4 (N = 38) | 4.68 (11.81)
  Week 8 (N = 36) | 2.06 (5.79)
  Week 12 (N = 36) | 1.81 (6.15)
  Week 24 (N = 36) | 1.89 (6.89)
  Week 36 (N = 35) | 2.03 (5.70)
  Week 48 (N = 34) | 1.32 (3.76)
  Week 60 (N = 33) | 0.97 (2.98)
  Week 72 (N = 32) | 0.56 (1.29)
  Week 84 (N = 31) | 0.77 (2.00)
  Week 96 (N = 30) | 0.33 (1.03)

59. Other Pre Specified Outcome: Overall Back Pain Score for ERA Sub-population
Description: Overall back pain assessed by participant's parent using a 100 millimeter (mm) VAS with 0 mm= no pain and 100 mm= most severe pain.
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Etanercept
Number analyzed (Participants) | 38
mm
  Baseline (N = 37) | 25.94 (28.00)
  Week 4 (N = 38) | 14.24 (19.87)
  Week 8 (N = 36) | 12.94 (22.60)
  Week 12 (N = 36) | 11.83 (18.22)
  Week 24 (N = 36) | 9.81 (17.23)
  Week 36 (N = 35) | 10.16 (19.20)
  Week 48 (N = 34) | 8.62 (15.76)
  Week 60 (N = 32) | 5.13 (12.28)
  Week 72 (N = 32) | 6.03 (14.67)
  Week 84 (N = 31) | 5.03 (8.40)
  Week 96 (N = 30) | 2.37 (4.51)

60. Other Pre Specified Outcome: Nocturnal Back Pain Score for ERA Sub-population
Description: Nocturnal back pain assessed by participant's parent using a 100 mm VAS with 0 mm = no pain and 100 mm = most severe pain.
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Etanercept
Number analyzed (Participants) | 38
mm
  Baseline (N = 38) | 16.37 (27.76)
  Week 4 (N = 38) | 8.58 (19.31)
  Week 8 (N = 36) | 7.82 (18.34)
  Week 12 (N = 36) | 5.81 (11.74)
  Week 24 (N = 36) | 5.31 (15.17)
  Week 36 (N = 35) | 7.54 (17.66)
  Week 48 (N = 34) | 5.85 (13.82)
  Week 60 (N = 32) | 3.34 (13.36)
  Week 72 (N = 32) | 6.47 (19.64)
  Week 84 (N = 31) | 2.66 (6.86)
  Week 96 (N = 30) | 2.17 (3.50)

61. Other Pre Specified Outcome: Modified Schober's Test for ERA Sub-population
Description: Modified Schober's Test: A mark was placed in the midpoint of a line that joined the posterior superior iliac spines. Another mark was placed 10 centimeter (cm) above the first. The participant then bent maximally forward with the knees fully extended. The distance between the two marks was then re-measured. The full measurement between the two lines was recorded to the nearest tenth of a centimeter.
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Etanercept
Number analyzed (Participants) | 127
cm
  Baseline (N = 37) | 5.03 (1.94)
  Week 4 (N = 38) | 5.24 (1.94)
  Week 8 (N = 36) | 5.12 (2.36)
  Week 12 (N = 36) | 5.45 (1.98)
  Week 24 (N = 36) | 5.35 (2.10)
  Week 36 (N = 35) | 5.49 (2.10)
  Week 48 (N = 34) | 5.38 (1.59)
  Week 60 (N = 33) | 5.33 (1.71)
  Week 72 (N = 32) | 5.27 (1.59)
  Week 84 (N = 30) | 5.47 (1.68)
  Week 96 (N = 30) | 5.33 (1.65)

62. Other Pre Specified Outcome: Percentage of Body Surface Area (BSA) Affected by Psoriasis for PsA Sub-population
Description: Percentage of body surface area affected by psoriasis was estimated using the palm method: one of the participant's palm to proximal interphalangeal and thumb= 1 percent (%) of BSA. Regions of the body were assigned specific number of palms with percentage [Head and neck= 10% (10 palms), upper extremities= 20% (20 palms), Trunk (axillae and groin)= 30% (30 palms), lower extremities (buttocks)= 40% (40 palms)]. The total BSA affected was the summation of individual regions affected.
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percentage of BSA
Arm/Group | Etanercept
Number analyzed (Participants) | 29
Percentage of BSA
  Baseline (N = 29) | 9.83 (13.61)
  Week 4 (N = 29) | 6.81 (9.02)
  Week 8 (N = 29) | 4.67 (7.68)
  Week 12 (N = 29) | 3.49 (5.66)
  Week 24 (N = 28) | 2.36 (4.24)
  Week 36 (N = 28) | 2.91 (8.70)
  Week 48 (N = 28) | 3.12 (8.13)
  Week 60 (N = 27) | 1.48 (2.38)
  Week 72 (N = 27) | 1.53 (2.17)
  Week 84 (N = 27) | 1.56 (2.27)
  Week 96 (N = 25) | 1.14 (2.12)

63. Other Pre Specified Outcome: Physician's Global Assessment (PGA) of Psoriasis for PsA Sub-population
Description: PGA of Psoriasis assessed the amount of induration, erythema, and scaling averaged over all psoriatic lesions on a scale of 0 to 5. 0 (no psoriasis) to 5 (severe disease). 'Clear' and "Almost clear' includes all participants who were scored as a 0 or 1.
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 29
Units on a scale
  Baseline (N = 29) | 1.76 (1.46)
  Week 4 (N = 29) | 1.41 (1.18)
  Week 8 (N = 29) | 1.07 (1.03)
  Week 12 (N = 28) | 0.82 (0.72)
  Week 24 (N = 28) | 0.61 (0.69)
  Week 36 (N = 28) | 0.61 (0.88)
  Week 48 (N = 28) | 0.75 (0.89)
  Week 60 (N = 27) | 0.78 (0.97)
  Week 72 (N = 26) | 0.65 (0.94)
  Week 84 (N = 27) | 0.56 (0.85)
  Week 96 (N = 25) | 0.48 (0.82)

64. Other Pre Specified Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. Number of participants reporting adverse events included medically important infections, infections considered preventable by vaccination, injection site reactions (ISRS), malignancies, adverse events, excluding infections and injection site reactions, infections and serious adverse events including infections.
Time Frame: Week 12, Week 96
Population: Safety population included all participants who received at least 1 dose of the study medication. Data are presented for Part 1 (up to 12 weeks) and Part 2 (up to 96 weeks).
Measure: Number; unit: Participants
Arm/Group | Etanercept
Number analyzed (Participants) | 127
Participants
  Medically important infections | 11
  Vaccine preventable infections | 8
  ISRs | 16
  Malignancies | 0
  Infections | 96
  Infection and ISRs excluded | 93
  Serious AE: Infection | 11

65. Other Pre Specified Outcome: Number of Participants With Adverse Events (AEs): eoJIA Subpopulation
Description: as for outcome 64
Time Frame: Week 12, Week 96
Population: as for outcome 23
Measure: Number; unit: Participants
Arm/Group | Etanercept
Number analyzed (Participants) | 60
Participants
  Medically important infections | 4
  Vaccine preventable infections | 6
  ISRs | 8
  Malignancies | 0
  Infections | 48
  Infection and ISRs excluded | 44
  Serious AE: Infection | 4

66. Other Pre Specified Outcome: Number of Participants With Adverse Events (AEs): ERA Sub-population
Description: as for outcome 64
Time Frame: Week 12, Week 96
Population: ERA:participants with Ar/enthesitis, any 2: sacroiliac joint tenderness/Ifm lumbosacral pain history; ankylosing spondylitis, ERA, sacroiliitis with Ifm bowel disease, Reiter's syndrome history; human leukocyte antigen-B27;Ar in male>6yrs; AAU/AAU in first-degree relative. Data are presented for Part 1 (up to 12 weeks) and Part 2 (up to 96 weeks).
Measure: Number; unit: Participants
Arm/Group | Etanercept
Number analyzed (Participants) | 38
Participants
  Medically important infections | 4
  Vaccine preventable infections | 1
  ISRs | 6
  Malignancies | 0
  Infections | 28
  Infection and ISRs excluded | 30
  Serious AE: Infection | 4

67. Other Pre Specified Outcome: Number of Participants With Adverse Events (AEs): PsA Sub-population
Description: as for outcome 64
Time Frame: Week 12, Week 96
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Etanercept
Number analyzed (Participants) | 29
Participants
  Medically important infections | 3
  Vaccine preventable infections | 1
  ISRs | 2
  Malignancies | 0
  Infections | 20
  Infection and ISRs excluded | 19
  Serious AE: Infection | 3

68. Other Pre Specified Outcome: Tanner Assessment Score by Age Group
Description: Tanner assessment score: used to document the stage of development of secondary sexual characteristics. Female pubertal development staged by pubic hair development and breast size; male pubertal development staged by size of the genitalia and development of pubic hair. Rated in 5 stages: stage 1 (no development) to 5 (adult-like development in quantity and size).
Time Frame: Baseline, Week 12, Week 48, Week 96
Population: Safety population: participants who received at least 1 dose of study medication. Data are presented for Part 1 (up to 12 weeks) and Part 2 (up to 96 weeks).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 127
Units on a scale
  Baseline: 2 to 17 years (N = 126) | 3.08 (1.59)
  Week 12: 2 to 17 years (N = 122) | 3.18 (1.63)
  Week 48: 2 to 17 years (N = 118) | 3.34 (1.61)
  Week 96: 2 to 17 years (N = 106) | 3.57 (1.61)

69. Other Pre Specified Outcome: Tanner Assessment Score by Age Group for eoJIA Sub-population
Description: as for outcome 68
Time Frame: Baseline, Week 12, Week 48, Week 96
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 60
Units on a scale
  Baseline: 2 to 4 years (N=14) | 1.00 (0.00)
  Baseline: 5 to 11 years (N=23) | 1.16 (0.44)
  Baseline: 12 to 17 years (N=22) | 3.94 (0.97)
  Baseline: 2 to 17 years (N=59) | 2.16 (1.53)
  Week 12: 2 to 4 years (N=14) | 1.00 (0.00)
  Week 12: 5 to 11 years (N=22) | 1.17 (0.45)
  Week 12: 12 to 17 years (N=21) | 4.02 (0.95)
  Week 12: 2 to 17 years (N=57) | 2.18 (1.56)
  Week 48: 2 to 4 years (n=13) | 1.00 (0.00)
  Week 48: 5 to 11 years (N=22) | 1.30 (0.63)
  Week 48: 12 to 17 years (N=21) | 4.35 (0.83)
  Week 48: 2 to 17 years (N=56) | 2.37 (1.67)
  Week 96: 2 to 4 years (N=13) | 1.00 (0.00)
  Week 96: 5 to 11 years (N=19) | 1.67 (1.08)
  Week 96: 12 to 17 years (N=20) | 4.53 (0.62)
  Week 96: 2 to 17 years (N=52) | 2.60 (1.73)

70. Other Pre Specified Outcome: Tanner Assessment Score by Age Group for ERA Sub-population
Description: as for outcome 68
Time Frame: Baseline, Week 12, Week 48, Week 96
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 38
Units on a scale
  Baseline: 12 to 17 years (N = 38) | 3.87 (1.07)
  Week 12: 12 to 17 years (N = 36) | 4.09 (1.04)
  Week 48: 12 to 17 years (N = 34) | 4.24 (0.84)
  Week 96: 12 to 17 years (N = 30) | 4.51 (0.66)

71. Other Pre Specified Outcome: Tanner Assessment Score by Age Group for PsA Sub-population
Description: as for outcome 68
Time Frame: Baseline, Week 12, Week 48, Week 96
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 29
Units on a scale
  Baseline: 12 to 17 years (N = 29) | 3.93 (1.22)
  Week 12: 12 to 17 years (N = 29) | 4.02 (1.19)
  Week 48: 12 to 17 years (N = 28) | 4.20 (0.95)
  Week 96: 12 to 17 years (N = 24) | 4.51 (0.69)

72. Other Pre Specified Outcome: Height z-Score by Age Group
Description: Standing height was taken as a mean of 3 consecutive measurements using a wall mounted stadiometer. Z-Score was a statistical measure to evaluate how a single data point compares to a standard. It described whether a mean was above or below the standard and how unusual the measurement is with range from -3 to +3; 0 =same mean, >0 a greater mean, and <0 a lesser mean than the standard. Growth parameters were compared to a standard defined by Centers for Disease Control's growth charts.
Time Frame: Baseline, Week 12, Week 48, Week 72, Week 96
Population: as for outcome 68
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Etanercept
Number analyzed (Participants) | 127
z-score
  Baseline: 2 to 17 years (N = 125) | 0.19 (1.07)
  Week 12: 2 to 17 years (N = 123) | 0.31 (0.98)
  Week 48: 2 to 17 years (N = 118) | 0.34 (1.02)
  Week 72: 2 to 17 years (N = 114) | 0.41 (0.97)
  Week 96: 2 to 17 years (N = 109) | 0.39 (0.99)

73. Other Pre Specified Outcome: Height z-Score by Age Group for eoJIA Sub-population
Description: as for outcome 72
Time Frame: Baseline, Week 12, Week 48, Week 72, Week 96
Population: eoJIA sub-population: participants with arthritis affecting 1 to 4 joints during the first 6 months of the disease and had progressed to affect more than 4 joints after the first 6 months of disease. Data are presented for Part 1 (up to 12 weeks) and Part 2 (up to 96 weeks).
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Etanercept
Number analyzed (Participants) | 60
z-score
  Baseline: 2 to 4 years (N=15) | -0.24 (1.32)
  Baseline: 5 to 11 years (N=22) | 0.20 (1.35)
  Baseline: 12 to 17 years (N=21) | 0.13 (0.84)
  Baseline: 2 to 17 years (N=58) | 0.06 (1.17)
  Week 12: 2 to 4 years (N=15) | 0.17 (0.97)
  Week 12: 5 to 11 years (N=22) | 0.28 (1.23)
  Week 12: 12 to 17 years (N=21) | 0.16 (0.83)
  Week 12: 2 to 17 years (N=58) | 0.21 (1.02)
  Week 48: 2 to 4 years (N=14) | 0.37 (1.06)
  Week 48: 5 to 11 years (N=21) | 0.30 (1.30)
  Week 48: 12 to 17 years (N=21) | 0.18 (0.87)
  Week 48: 2 to 17 years (N=56) | 0.27 (1.08)
  Week 72: 2 to 4 years (N=14) | 0.39 (0.99)
  Week 72: 5 to 11 years (N=21) | 0.43 (1.11)
  Week 72: 12 to 17 years (N=20) | 0.20 (0.87)
  Week 72: 2 to 17 years (N=55) | 0.34 (0.98)
  Week 96: 2 to 4 years (N=14) | 0.34 (0.99)
  Week 96: 5 to 11 years (N=20) | 0.46 (1.15)
  Week 96: 12 to 17 years (N=20) | 0.17 (0.89)
  Week 96: 2 to 17 years (N=54) | 0.32 (1.01)

74. Other Pre Specified Outcome: Height z-Score by Age Group for ERA Sub-population
Description: as for outcome 72
Time Frame: Baseline, Week 12, Week 48, Week 72, Week 96
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Etanercept
Number analyzed (Participants) | 38
z-score
  Baseline: 12 to 17 years (N = 38) | 0.24 (0.89)
  Week 12: 12 to 17 years (N = 36) | 0.35 (0.86)
  Week 48: 12 to 17 years (N = 34) | 0.36 (0.85)
  Week 72: 12 to 17 years (N = 32) | 0.46 (0.84)
  Week 96: 12 to 17 years (N = 30) | 0.43 (0.86)

75. Other Pre Specified Outcome: Height z-Score by Age Group for PsA Sub-population
Description: as for outcome 72
Time Frame: Baseline, Week 12, Week 48, Week 72, Week 96
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Etanercept
Number analyzed (Participants) | 29
z-score
  Baseline: 12 to 17 years (N = 29) | 0.41 (1.06)
  Week 12: 12 to 17 years (N = 29) | 0.46 (1.05)
  Week 48: 12 to 17 years (N = 28) | 0.47 (1.11)
  Week 72: 12 to 17 years (N = 27) | 0.51 (1.10)
  Week 96: 12 to 17 years (N = 25) | 0.48 (1.11)

76. Other Pre Specified Outcome: Weight z-Scores by Age Group
Description: Weight was taken as a mean of 3 consecutive measurements using a medical electronic scale. Z-Score was a statistical measure to evaluate how a single data point compares to a standard. It described whether a mean was above or below the standard and how unusual the measurement is with range from -3 to +3; 0 =same mean, >0 a greater mean, and <0 a lesser mean than the standard. Growth parameters were compared to a standard defined by Centers for Disease Control's growth charts.
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: as for outcome 68
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Etanercept
Number analyzed (Participants) | 127
z-score
  Baseline: 2 to 17 years (N = 127) | 0.17 (1.02)
  Week 4: 2 to 17 years (N = 126) | 0.18 (1.02)
  Week 8: 2 to 17 years (N = 121) | 0.23 (1.02)
  Week 12: 2 to 17 years (N = 123) | 0.22 (1.00)
  Week 24: 2 to 17 years (N = 122) | 0.25 (0.99)
  Week 36: 2 to 17 years (N = 120) | 0.26 (0.97)
  Week 48: 2 to 17 years (N = 118) | 0.25 (0.97)
  Week 60: 2 to 17 years (N = 116) | 0.24 (0.95)
  Week 72: 2 to 17 years (N = 114) | 0.29 (0.91)
  Week 84: 2 to 17 years (N = 113) | 0.27 (0.93)
  Week 96: 2 to 17 years (N = 109) | 0.25 (0.93)

77. Other Pre Specified Outcome: Weight z-Scores by Age Group for eoJIA Sub-population
Description: as for outcome 76
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Etanercept
Number analyzed (Participants) | 60
z-score
  Baseline: 2 to 4 years (N=15) | -0.50 (0.98)
  Baseline: 5 to 11 years (N=23) | 0.15 (1.33)
  Baseline: 12 to 17 years (N=22) | 0.40 (0.72)
  Baseline: 2 to 17 years (N=60) | 0.08 (1.10)
  Week 4: 2 to 4 years (N=15) | -0.54 (1.13)
  Week 4: 5 to 11 years (N=23) | 0.17 (1.34)
  Week 4: 12 to 17 years (N=21) | 0.38 (0.69)
  Week 4: 2 to 17 years (N=59) | 0.06 (1.13)
  Week 8: 2 to 4 years (N=14) | -0.48 (1.25)
  Week 8: 5 to 11 years (N=21) | 0.30 (1.30)
  Week 8: 12 to 17 years (N=21) | 0.40 (0.72)
  Week 8: 2 to 17 years (N=56) | 0.14 (1.14)
  Week 12: 2 to 4 years (n=15) | -0.35 (1.09)
  Week 12: 5 to 11 years (N=22) | 0.22 (1.35)
  Week 12: 12 to 17 years (N=21) | 0.41 (0.72)
  Week 12: 2 to 17 years (N=58) | 0.14 (1.11)
  Week 24: 2 to 4 years (N=15) | -0.21 (1.10)
  Week 24: 5 to 11 years (N=22) | 0.21 (1.32)
  Week 24: 12 to 17 years (N=21) | 0.46 (0.69)
  Week 24: 2 to 17 years (N=58) | 0.19 (1.08)
  Week 36: 2 to 4 years (N=14) | -0.25 (1.14)
  Week 36: 5 to 11 years (N=22) | 0.27 (1.25)
  Week 36: 12 to 17 years (N=21) | 0.39 (0.70)
  Week 36: 2 to 17 years (N=57) | 0.18 (1.06)
  Week 48: 2 to 4 years (N=14) | -0.28 (1.15)
  Week 48: 5 to 11 years (N=21) | 0.21 (1.24)
  Week 48: 12 to 17 years (N=21) | 0.40 (0.65)
  Week 48: 2 to 17 years (N=56) | 0.16 (1.05)
  Week 60: 2 to 4 years (N=14) | -0.18 (1.15)
  Week 60: 5 to 11 years (N=22) | 0.23 (1.24)
  Week 60: 12 to 17 years (N=20) | 0.31 (0.62)
  Week 60: 2 to 17 years (N=56) | 0.16 (1.04)
  Week 72: 2 to 4 years (N=14) | -0.09 (1.12)
  Week 72: 5 to 11 years (N=21) | 0.43 (1.13)
  Week 72: 12 to 17 years (N=20) | 0.29 (0.67)
  Week 72: 2 to 17 years (N=55) | 0.25 (0.99)
  Week 84: 2 to 4 years (N=14) | -0.10 (1.13)
  Week 84: 5 to 11 years (N=21) | 0.42 (1.15)
  Week 84: 12 to 17 years (N=20) | 0.23 (0.74)
  Week 84: 2 to 17 years (N=55) | 0.22 (1.02)
  Week 96: 2 to 4 years (N=14) | -0.14 (1.18)
  Week 96: 5 to 11 years (N=20) | 0.49 (1.11)
  Week 96: 12 to 17 years (N=20) | 0.16 (0.76)
  Week 96: 2 to 17 years (N=54) | 0.20 (1.03)

78. Other Pre Specified Outcome: Weight z-Scores by Age Group for ERA Sub-population
Description: as for outcome 76
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Etanercept
Number analyzed (Participants) | 38
z-score
  Baseline: 12 to 17 years (N = 38) | -0.05 (0.74)
  Week 4: 12 to 17 years (N = 38) | -0.00 (0.72)
  Week 8: 12 to 17 years (N = 36) | 0.04 (0.68)
  Week 12: 12 to 17 years (N = 36) | -0.00 (0.65)
  Week 24: 12 to 17 years (N = 36) | 0.01 (0.68)
  Week 36: 12 to 17 years (N = 35) | 0.03 (0.68)
  Week 48: 12 to 17 years (N = 34) | 0.04 (0.70)
  Week 60: 12 to 17 years (N = 33) | 0.08 (0.67)
  Week 72: 12 to 17 years (N = 32) | 0.12 (0.65)
  Week 84: 12 to 17 years (N = 31) | 0.07 (0.67)
  Week 96: 12 to 17 years (N = 30) | 0.06 (0.63)

79. Other Pre Specified Outcome: Weight z-Scores by Age Group for PsA Sub-population
Description: as for outcome 76
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Etanercept
Number analyzed (Participants) | 29
z-score
  Baseline: 12 to 17 years (N = 29) | 0.63 (1.05)
  Week 4: 12 to 17 years (N = 29) | 0.66 (1.01)
  Week 8: 12 to 17 years (N = 29) | 0.64 (1.04)
  Week 12: 12 to 17 years (N = 29) | 0.63 (1.04)
  Week 24: 12 to 17 years (N = 28) | 0.66 (1.04)
  Week 36: 12 to 17 years (N = 28) | 0.69 (0.97)
  Week 48: 12 to 17 years (N = 28) | 0.70 (0.96)
  Week 60: 12 to 17 years (N = 27) | 0.61 (1.00)
  Week 72: 12 to 17 years (N = 27) | 0.57 (0.97)
  Week 84: 12 to 17 years (N = 27) | 0.59 (0.94)
  Week 96: 12 to 17 years (N = 25) | 0.59 (0.96)

80. Other Pre Specified Outcome: Body Mass Index (BMI) z-Score by Age Group
Description: BMI was used to measure body fat based on height and weight. It was calculated by body weight (kg)/height (m) squared. Z-Score was a statistical measure to evaluate how a single data point compares to a standard. It described whether a mean was above or below the standard and how unusual the measurement is with range from -3 to +3; 0 =same mean, >0 a greater mean, and <0 a lesser mean than the standard. Growth parameters were compared to a standard defined by Centers for Disease Control's growth charts.
Time Frame: Baseline, Week 12, Week 48, Week 72, Week 96
Population: as for outcome 68
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Etanercept
Number analyzed (Participants) | 127
z-score
  Baseline: 2 to 17 years (N = 125) | 0.03 (1.17)
  Week 12: 2 to 17 years (N = 123) | 0.03 (1.15)
  Week 48: 2 to 17 years (N = 118) | 0.05 (1.11)
  Week 72: 2 to 17 years (N = 114) | 0.07 (1.03)
  Week 96: 2 to 17 years (N = 109) | 0.04 (1.06)

81. Other Pre Specified Outcome: Body Mass Index (BMI) z-Score by Age Group for eoJIA Sub-population
Description: as for outcome 80
Time Frame: Baseline, Week 12, Week 48, Week 72, Week 96
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Etanercept
Number analyzed (Participants) | 60
z-score
  Baseline: 2 to 4 years (N=15) | -0.60 (1.70)
  Baseline: 5 to 11 years (N=22) | 0.03 (1.28)
  Baseline: 12 to 17 years (N=21) | 0.40 (0.72)
  Baseline: 2 to 17 years (N=58) | 0.00 (1.28)
  Week 12: 2 to 4 years (N=15) | -0.78 (1.64)
  Week 12: 5 to 11 years (N=22) | 0.21 (1.13)
  Week 12: 12 to 17 years (N=21) | 0.38 (0.73)
  Week 12: 2 to 17 years (N=58) | 0.01 (1.25)
  Week 48: 2 to 4 years (N=14) | -0.85 (1.69)
  Week 48: 5 to 11 years (N=21) | 0.18 (0.96)
  Week 48: 12 to 17 years (N=21) | 0.34 (0.68)
  Week 48: 2 to 17 years (N=56) | -0.02 (1.19)
  Week 72: 2 to 4 years (N=14) | -0.48 (1.46)
  Week 72: 5 to 11 years (N=21) | 0.37 (0.97)
  Week 72: 12 to 17 years (N=20) | 0.20 (0.73)
  Week 72: 2 to 17 years (N=55) | 0.09 (1.08)
  Week 96: 2 to 4 years (N=14) | -0.50 (1.55)
  Week 96: 5 to 11 years (N=20) | 0.44 (0.90)
  Week 96: 12 to 17 years (N=20) | 0.05 (0.83)
  Week 96: 2 to 17 years (N=54) | 0.05 (1.13)

82. Other Pre Specified Outcome: Body Mass Index (BMI) z-Score by Age Group for ERA Sub-population
Description: as for outcome 80
Time Frame: Baseline, Week 12, Week 48, Week 72, Week 96
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Etanercept
Number analyzed (Participants) | 38
z-score
  Baseline: 12 to 17 years (N = 38) | -0.29 (0.87)
  Week 12: 12 to 17 years (N = 36) | -0.31 (0.86)
  Week 48: 12 to 17 years (N = 34) | -0.27 (0.91)
  Week 72: 12 to 17 years (N = 32) | -0.23 (0.87)
  Week 96: 12 to 17 years (N = 30) | -0.29 (0.84)

83. Other Pre Specified Outcome: Body Mass Index (BMI) z-Score by Age Group for PsA Sub-population
Description: as for outcome 80
Time Frame: Baseline, Week 12, Week 48, Week 72, Week 96
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Etanercept
Number analyzed (Participants) | 29
z-score
  Baseline: 12 to 17 years (N = 29) | 0.51 (1.17)
  Week 12: 12 to 17 years (N = 29) | 0.49 (1.14)
  Week 48: 12 to 17 years (N = 28) | 0.55 (1.01)
  Week 72: 12 to 17 years (N = 27) | 0.37 (1.04)
  Week 96: 12 to 17 years (N = 25) | 0.40 (1.06)

84. Other Pre Specified Outcome: Number of Participants With Anti-etanercept Antibodies
Time Frame: Baseline up to Week 12, Week 48, Week 96
Population: as for outcome 64
Measure: Number; unit: Participants
Arm/Group | Etanercept
Number analyzed (Participants) | 127
Participants
  Overall (N=127) | 26
  Week 12 (N=120) | 6
  Week 48 (N=116) | 14
  Week 96 (N=105) | 14

85. Other Pre Specified Outcome: Number of Participants With Anti-etanercept Antibodies: eoJIA Sub-population
Time Frame: Baseline up to Week 12, Week 48, Week 96
Population: as for outcome 23
Measure: Number; unit: Participants
Arm/Group | Etanercept
Number analyzed (Participants) | 60
Participants
  Overall (N=60) | 11
  Week 12 (N=56) | 0
  Week 48 (N=55) | 7
  Week 96 (N=52) | 7

86. Other Pre Specified Outcome: Number of Participants With Anti-etanercept Antibodies: ERA Sub-population
Time Frame: Baseline up to Week 12, Week 48, Week 96
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | Etanercept
Number analyzed (Participants) | 38
Participants
  Overall (N=38) | 9
  Week 12 (N=36) | 4
  Week 48 (N=34) | 4
  Week 96 (N=29) | 3

87. Other Pre Specified Outcome: Number of Participants With Anti-etanercept Antibodies: PsA Sub-population
Time Frame: Baseline up to Week 12, Week 48, Week 96
Population: PsA: participants with arthritis and psoriasis, or arthritis plus at least 2 of the following: 1) dactylitis; 2) nail pitting or onycholysis; 3) psoriasis in a firstdegree relative. Data are presented for Part 1 (up to 12 weeks) and Part 2 (up to 96 weeks).
Measure: Number; unit: Participants
Arm/Group | Etanercept
Number analyzed (Participants) | 29
Participants
  Overall (N=29) | 6
  Week 12 (N=28) | 2
  Week 48 (N=27) | 3
  Week 96 (N=24) | 4

88. Other Pre Specified Outcome: Number of Participants With Neutralizing Anti-etanercept Antibodies
Time Frame: Baseline up to Week 12, Week 48, Week 96
Population: Safety population included all participants who received at least 1 dose of the study medication.
Measure: Number; unit: Participants
Arm/Group | Etanercept
Number analyzed (Participants) | 127
Participants | 0

ADVERSE EVENTS:
Time Frame: Screening up to Week 96
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Etanercept
Serious Adverse Events (participants affected / at risk) | 24/127
Other Adverse Events (participants affected / at risk) | 106/127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (N=127)
Abdominal pain (Gastrointestinal disorders) | 1
Bronchopneumonia (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 2
Pyelocystitis (Infections and infestations) | 1
Phimosis (Congenital, familial and genetic disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Crohn's disease (Gastrointestinal disorders) | 1
Acute tonsillitis (Infections and infestations) | 1
Gastrointestinal infection (Infections and infestations) | 1
Helicobacter gastritis (Infections and infestations) | 1
Peritonitis (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Cartilage injury (Injury, poisoning and procedural complications) | 1
Concussion (Injury, poisoning and procedural complications) | 1
Forearm fracture (Injury, poisoning and procedural complications) | 1
Fractured coccyx (Injury, poisoning and procedural complications) | 1
Tendon injury (Injury, poisoning and procedural complications) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Juvenile arthritis (Musculoskeletal and connective tissue disorders) | 2
Syncope (Nervous system disorders) | 1
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1
Adenoidectomy (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (N=127)
Abdominal pain (Gastrointestinal disorders) | 6
Diarrhoea (Gastrointestinal disorders) | 10
Pyrexia (General disorders) | 9
Bronchitis (Infections and infestations) | 13
Gastroenteritis (Infections and infestations) | 18
Nasopharyngitis (Infections and infestations) | 16
Pharyngitis (Infections and infestations) | 32
Rhinitis (Infections and infestations) | 11
Upper respiratory tract infection (Infections and infestations) | 42
Headache (Nervous system disorders) | 17
Anaemia (Blood and lymphatic system disorders) | 4
Leukopenia (Blood and lymphatic system disorders) | 7
Neutropenia (Blood and lymphatic system disorders) | 4
Conjunctivitis (Eye disorders) | 5
Gastritis (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 5
Influenza like illness (General disorders) | 11
Ear infection (Infections and infestations) | 9
Sinusitis (Infections and infestations) | 6
Tonsillitis (Infections and infestations) | 9
Alanine aminotransferase increased (Investigations) | 6
Aspartate aminotransferase increased (Investigations) | 6
Hepatic enzyme increased (Investigations) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 6
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 4

LIMITATIONS AND CAVEATS:
Results include data for Part 1 (up to Week 12) and Part 2 (up to week 96) of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.